CLINICAL TRIAL: NCT06847763
Title: The Effect of Online Therapeutic Neuroscience Education Added to Conventional Physiotherapy Program on Clinical Outcomes, Treatment Expectations and Satisfaction Levels in Patients With Chronic Low Back Pain
Brief Title: The Long Term Effects of Online Therapeutic Neuroscience Education in Patients With Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulBUFC8
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain, Mechanical; Chronic Pain
Keywords: therapeutic neuroscience education; chronic low back pain; kinesiophobia; disability; treatment expectation
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): These participants will receive online Therapeutic Neuroscience Education with conventional physiotherapy program.
  Interventions: Other: Therapeutic Neuroscience Education; Other: Conventional Program
- Control (Active Comparator): Control group will receive only conventional physiotherapy program.
  Interventions: Other: Conventional Program

INTERVENTIONS:
Other: Therapeutic Neuroscience Education — Therapeutic Neuroscience Education applied in the form of one-on-one seminar format, focused on pain neurophysiology, and in the form of speaking sessions. Within the scope of these speaking sessions, pictures, diagrams, graphs, examples, metaphors, and homework assignments explaining the neurophysiology of pain are used.
  Arms: Experimental
Other: Conventional Program — Conventional physiotherapy includes hot packs (20 minutes), ultrasound (1 mHz frequency, 1,5 watt/cm², 5 minutes left/right lumbar region), TENS (100Hz, 20 minutes), and home exercises.

SUMMARY:
This study aims to evaluate the effects of online Therapeutic Neuroscience Education (TNE) combined with a 6-week conventional physiotherapy program on pain, disability, kinesiophobia, functionality, treatment expectations, and satisfaction in individuals with chronic low back pain (CLBP). The goal is to improve participants' understanding of chronic pain, reduce fear and avoidance behaviors, enhance movement and functionality, and increase treatment satisfaction. The study also seeks to provide a lasting educational resource.

TNE focuses on educating patients about pain neurophysiology, aiming to reduce pain, improve function, and shift perceptions about pain through interactive sessions involving diagrams, metaphors, and examples. Despite evidence supporting TNE's effectiveness for chronic pain conditions, no studies have evaluated its online application or long-term effects.

The study will include 60 volunteers with CLBP (ages 20-60), randomized into two groups: one receiving conventional physiotherapy and online TNE, and the other receiving conventional treatment alone. The TNE group will participate in six weekly 45-minute online sessions, covering topics like pain neurophysiology, biopsychosocial factors, and pain coping strategies, without addressing anatomical or emotional aspects.

Educational materials, including resources adapted from "Why You Hurt" will be presented to the TNE group. Conventional physiotherapy includes hot packs, ultrasound, TENS, and home exercises for both groups.

Clinical outcomes will be assessed by a blinded researcher at multiple time points using tools such as pain and disability scales, kinesiophobia measures, functional tests, and questionnaires on treatment expectations and satisfaction. The study is significant for its innovative approach in examining the clinical and long-term effectiveness of online TNE as part of CLBP management.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of therapeutic neuroscience education applied online in addition to a 6-week conventional physiotherapy program on pain, disability, kinesiophobia, functionality, treatment expectations and satisfaction in individuals with chronic low back pain.

At the end of the study, it is aimed to help individuals with chronic low back pain better understand the biological process underlying chronic pain conditions with therapeutic neuroscience education; to increase treatment expectations and satisfaction by achieving therapeutic effects such as reducing fear associated with pain and musculoskeletal injuries, and increasing movement and functionality.

In individuals with chronic low back pain, the disease state, fear and avoidance behavior related to the treatment process, catastrophizing, inappropriate beliefs and psychosocial factors (yellow flags) cause pain to increase and become chronic.

Therapeutic Neuroscience Education (TNE) is an information application applied by a physiotherapist with therapeutic purposes such as reducing pain, improving function, helping the individual understand the cause of their pain, and reconceptualizing pain. It is used to raise awareness about pain and the coding of pain in the brain, to improve the individual's health behavior and health status, and to stimulate the cognitive infrastructure. TNE is a method applied in the form of one-on-one seminar format, focused on pain neurophysiology, and in the form of speaking sessions. Within the scope of these speaking sessions, pictures, diagrams, graphs, examples, metaphors, and homework assignments explaining the neurophysiology of pain are used.

There are findings that Therapeutic Neuroscience Education improves pain and disability in various populations with chronic pain (such as low back/neck pain, fibromyalgia), but there is no protocol in the literature showing the effectiveness of the TNE program given online.

The importance of this study is that it will be an innovative study examining the effectiveness of online TNE, in addition to conventional physiotherapy programs, on clinical outcomes in individuals with chronic low back pain, as well as individuals' treatment expectations and satisfaction.

60 volunteers with chronic low back pain between the ages of 20-60 will be included in the study. Participants will be randomly assigned to Online TNE (n=30) and Control (n=30) groups that will receive conventional treatment according to an internet-based randomization program.

The online training modules to be used in the first phase of the study will be structured specifically for individuals with chronic low back pain. The training program will be created in 6 sessions lasting 45 minutes in total and one session for a week.

Within the scope of TNE training; chronic pain, pain and injury are not equivalent, pain is an output produced in the brain rather than an input, biopsychosocial factors, neurophysiology of pain, nociception and nociceptive pathways, neurons, synapses, action potential, spinal inhibition and facilitation, sensitization, extra sensitive nerves and alarm system, stress, fear, avoidance and effects on pain, plasticity of the nervous system, pain coping strategies and effects of movement on chronic pain will be discussed with metaphors and stories. Anatomical and pathoanatomical models will not be addressed, and emotional or behavioral aspects of pain will not be included.

Participants in the TNE group will be presented with illustrated cards as training materials, including various examples, metaphors, and assignments developed to facilitate individual understanding.

In the second phase of the study, the effectiveness of the online education program will be evaluated. In addition to the conventional physiotherapy program, the TNE group will be provided with one session of therapeutic neuroscience education online for six weeks. The password-protected zoom platform will be used for online education. The conventional physiotherapy program will be given all participants and included hot pack, ultrasound, TENS and a standard home exercise program to strengthen the abdominal and back muscles.

The participants will be evaluated by an independent researcher at baseline, in the third week, at the 6th week and 6 months after the study in a blinded manner.

Participants' pain will be assessed with the Numeric Pain Scale and Pain Catastrophizing Scale, fear and anxiety related to movement with the Tampa Scale of Kinesiophobia, and disabilities with the Roland Morris Disability Questionnaire and Timed Up and Go Test. The flexibility of the lumbar extensors will be measured by the forward bending distance. Treatment Expectations will be assessed with the Treatment Expectation Questionnaire at the beginning and middle of the program, and treatment satisfaction will be assessed with the Patient Satisfaction Scale in Physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20-60
* Literate
* Having received a score of 24 or above in the Mini-Mental Status Assessment
* Having internet access
* Having back pain for more than 3 months
* Having pain between 3-8 on the Numerical Pain Scale
* Individuals with chronic back pain whose symptoms are not radicular

Exclusion Criteria:

* Having other orthopedic/neurological disorders that will affect the evaluation and treatment
* Patients with vertebral compression fractures on MRI and lumbar radiography
* Patients with unstable neurological findings
* Patients using analgesic medication during treatment
* Patients with rheumatological and inflammatory diseases
* Patients with acute trauma
* Patients who are pregnant
* Patients who have undergone lumbar region surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | T0 (baseline), T1 (3rd week), T2 (6th week) and T3 (6 month follow up)
  Tampa Scale of Kinesiophobia will be used to assess kinesiophobia, which is an anxiety state that develops against activity and physical movement. This scale was developed to distinguish between non-excessive fear and phobia in individuals with chronic musculoskeletal pain. It is widely used in the literature to assess fear and anxiety related to movement. The scale consists of 17 items covering work-related activities, injury, re-injury, and fear-avoidance parameters and scored between 17-68. High scores obtained from the scale indicate that the individual's level of kinesiophobia has increased. Studies conducted on patients with low back and neck pain have revealed that the test-retest reliability ICC value of the Turkish version of the scale is 0.80.
Pain Level | T0 (baseline), T1 (3rd week), T2 (6th week) and T3 (6 month follow up)
  Numeric Pain Scale will be used for assessing the participants' pain levels. Participants will be asked to determine the number that best describes their pain on a scale of 0 to 10, where 0 = no pain and 10 = unbearable pain. The Numerical Pain Scale is a valid and reliable measurement method for subjective pain intensity assessment. Rest, activity and night pain will be located on a horizontal stripe that the participant will mark. High numbers indicated higher pain levels.
Pain Catastrophizing | T0 (baseline), T1 (3rd week), T2 (6th week) and T3 (6 month follow up)
  The Pain Catastrophizing Scale will be used to assess participants' pain catastrophizing. This scale is a self-report questionnaire that assesses unhelpful coping strategies and catastrophizing thoughts about pain and injury and has strong validity and reliability. The scale consists of 13 questions, each question is scored between 0 and 4. The lowest possible score is 0, the highest score is 52. As the score increases (e.g. >10), pain catastrophizing thoughts increase. The Turkish validity and reliability study of the questionnaire was conducted and Cronbach's alpha value was reported as 0.955 and ICC value as 0.830.

SECONDARY OUTCOMES:
Disability | T0 (baseline), T1 (3rd week), T2 (6th week) and T3 (6 month follow up)
  The Roland Morris Disability Questionnaire will be used to determine the physical adequacy level of the participants. The questionnaire consists of 24 items and yes/no answers are given for each activity. A yes answer is scored as 1 point, a no answer as 0 points. The lowest score on this scale is 0, and the highest score is 24. High scores indicate inadequacy in physical activities. The Turkish validity and reliability study of the questionnaire was conducted and the Cronbach alpha internal consistency value was reported as over 0.85.
Physical Function | T0 (baseline), T1 (3rd week), T2 (6th week) and T3 (6 month follow up)
  The Timed Up and Go Test will be used to assess functional status. This performance test covers basic motor skills such as static balance, dynamic balance, mobility and turning. During the test, the individual will get up from a seated position, walk a distance of 3 meters, return and sit down again. The test duration will be measured in seconds and recorded.The validity and reliability of the test in individuals with chronic low back pain has been proven.
Treatment Expectation | T0 (baseline), T1 (3rd week)
  Participants' treatment expectation levels will be assessed with the Treatment Expectations Questionnaire. The questionnaire, consisting of 15 main items, is in the form of a scale where the individual marks his/her treatment expectation between 0 and 10. The cumulative score of the questionnaire is 150 and the internal consistency Cronbach's alpha value of the original version was reported as 0.79 and the test-retest reliability was high (0.76). The Turkish validity and reliability of the questionnaire was conducted and the internal consistency Cronbach's alpha value was reported as 0.832.
Treatment Satisfaction | T2 (6th week) and T3 (6 month follow up)
  Participants' treatment satisfaction will be evaluated with a subjective mini-survey in 5-point Likert form prepared by the researchers. Treatment satisfaction will be scored between 5-25.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Gulden Polat, Prof., Study Director — Marmara University
Locations (1):
- Ornek Medical Clinic, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No